CLINICAL TRIAL: NCT01749345
Title: Social Determinants of Health as Explanatory Factors for Ethnic Disparities in Diabetes Outcomes
Brief Title: Social Determinants of Health in Diabetes Outcomes
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17676; 1K24DK093699-01 (NIH)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
This is a cross-sectional study of six hundred adults with type 2 diabetes, (300 White and 300 African-American) who will be recruited from two primary care sites to determine how social determinants of health impact diabetes outcomes. The first aim is to investigate the role of psychosocial factors and SES on diabetes care processes and outcomes. The second aim is to investigate the influence of community and neighborhood characteristics on diabetes care processes and outcomes. Finally, we will examine the contribution of social determinants of health to ethnic differences in diabetes care processes and outcomes. Clinical and metabolic measures will be abstracted from the electronic medical records. Outcome variables include hemoglobin A1c, blood pressure, LDL-Cholesterol and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Able to communicate in English

Exclusion Criteria:

* Mental confusion on interview suggesting significant dementia
* Alcohol or drug abuse/dependency
* Active psychosis or acute mental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pimary care and internal medicine clinics
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
HbA1C | Within 3 months prior to the assessment
Quality of life | Within a month of completely the assessment

SECONDARY OUTCOMES:
Blood pressure | Most recent to assessment date
Low density lipoprotein (LDL) Cholesterol | Most recent to assessment date

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, M.D., Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina